CLINICAL TRIAL: NCT04248257
Title: Peer Support For Young Adult Women With High Breast Cancer Risk
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00001007
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PeACE peer coaching arm (Experimental): Behavioral, PeACE, PeACE consists of 3 streamlined 30-minute psychosocial telephone counseling sessions delivered by a well-trained peer coach. Coaches are lay YARs from HBOC families demonstrating good knowledge, communication skills, and protocol mastery.
  Interventions: Behavioral: PeACE
- Community peer coaching arm (Active Comparator): Behavioral, usual care, Participants in the usual care arm will receive navigation to peer support with a range of community groups who provide these services.
  Interventions: Behavioral: Community peer coaching

INTERVENTIONS:
Behavioral: PeACE — 3 session peer coaching intervention
  Arms: PeACE peer coaching arm
Behavioral: Community peer coaching — Peer coaching provided by community organizations that support the HBOC community
  Arms: Community peer coaching arm

SUMMARY:
This trial will recruit young adult female relatives (YARs) of male or female carriers of BRCA1/2. YARs who consent to participate will be randomized to either a 3-session peer coach-led telephone counseling intervention or usual care navigation to peer support interventions provided by community organizations that support the hereditary cancer community. Study aims are to 1) Assess intervention effects on distress and decision making outcomes, including uptake of counseling for untested YARs, 2) Identify YARs most likely to engage with and benefit from the intervention, 3) Understand intervention mechanisms. Participants will complete interviews at baseline, 1, 6, and 12 months.

DETAILED DESCRIPTION:
Germline (e.g., BRCA) mutation carriers have highly elevated odds of developing hereditary breast-ovarian cancer (HBOC), as could their relatives. Referral to genetic counseling is the standard of care for young, at-risk adult relatives (i.e., ages 18-39; herein "YARs"). However, many female YARs struggle to make decisions about familial HBOC risk management, including whether and when to pursue genetic counseling, how to cope with stress and uncertainty about HBOC, and how to navigate lifecycle events entwined with HBOC threats (e.g., childbearing). Prior work points to YARs' strong desires to seek HBOC risk information and emotional support beyond traditional genetic counseling-especially support from knowledgeable peers who can relate to their experiences and offer neutral grounding and objective guidance about coping strategies. Peer support is a promising psychosocial cancer care approach that could fill this void. However, few evidence-based standards inform its practice as an adjunct to cancer genetic counseling. As genetic testing for HBOC risk expands population-wide, new ways must be tested to reach, educate, and support YARs to further reduce the cancer burden in communities of at-risk women. The 2-arm PeACE trial includes streamlined telephone counseling delivered by well-trained community peer coaches, with session content incorporating coping training for HBOC stress reduction, and decision making and problem solving training about genetic counseling and HBOC risk. Trial participants are female YARs (aged 21-30) randomized to an intervention or equated control condition, and followed for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* There are two targets for recruitment with different eligibility criteria.

Index carriers:

* Men or women aged 18 or older with BRCA mutations with or without 2nd-tier multiplex panel genetic testing. Index carriers will have received testing.

YARs:

* Female 1st-, 2nd- or 3rd-degree biological relatives of index carriers aged 21-30.

Exclusion Criteria:

* Must be able to speak English or Spanish and provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Index carriers can be men and women; those taking part in peer coaching will be female.
Enrollment: 560 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cancer-related distress | 12 months
  Cancer-related distress about hereditary breast and ovarian cancer risk at 12 months, gathered via self-report using the Impact of Events Scale, a 15 item measure scored on a 0-3 scale (0-45) with higher scores meaning higher distress
Decisional conflict | 12 months
  Decisional conflict about hereditary breast and ovarian cancer risk management decisions at 12 months gathered via self-report using the Decisional Conflict Scale. The 16 items on a 0-4 scale are summed, divided by 16 and multiplied by 25 for a total score (range=0-100); higher scores indicate higher conflict
Genetic counseling | 12 months
  Genetic counseling uptake at 12 months gathered via self-report (for untested women); this is a binary yes/no question

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne O'Neill, Principal Investigator — Georgetown University
Locations (6):
- United States (6):
  - Georgetown University, Washington D.C., District of Columbia
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington